CLINICAL TRIAL: NCT06319092
Title: Validity and Reliability of an Immersive Virtual Reality Version of the 6 Minute Pegboard and Ring Test in Healthy Subjects
Brief Title: Immersive Virtual Reality Version of the 6 Minute Pegboard and Ring Test
Status: Completed | Type: Observational
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Çağtay Maden, Assistant professor, Gaziantep Islam Science and Technology University
Other Study IDs: 2023/175
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: 6 pegboard and ring test; upper extremity functional capacity; Healthy; handgrip

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The 6 Minute Pegboard and Ring Test is a test applicable to the upper extremities. The upper extremity plays an important role in activities of daily living, especially in tasks related to reaching, grasping and holding objects. Various activities of daily living, such as combing hair, brushing teeth and picking up objects, require supported or unsupported upper limb activity. Therefore, evaluation of upper extremity function is important. In addition, it is a simple test, it is also seen as a game, its application is functional, and there is no need for expensive equipment. Its validity and reliability have been demonstrated only for patients with Chronic Obstructive Pulmonary Disease (COPD) and healthy adults. In addition, to the best of our knowledge, the suitability of this test in a virtual environment has not been evaluated in the literature. Therefore, the main aim of this study is to examine the applicability of this test in a virtual environment.

DETAILED DESCRIPTION:
6 Minutes The virtual reality space for the Pegboard Ring Test will be designed in Blender programme. The software and integration that provides the interactive movement of the person in the application will be done by the UNITY programme.

Entry to the prepared training test area will be with OCULUS Quest 2 (virtual reality glasses and console) equipment.

ELIGIBILITY:
Inclusion Criteria:

* No orthopaedic problem or limitation of movement in the upper extremity that would adversely affect the test 6PBRT,
* no diagnosis or history of symptomatic lung and/or heart disease,
* no serious visual and hearing problems,
* no psychological and epileptic illnesses,
* not being diagnosed with migraine before,
* body mass index (BMI > 20.34, kg/m2 and < 25.94 kg/m2 for male individuals; BMI > 14.6 kg/m2 and < 25.55 kg/m2 for female individuals)

Exclusion Criteria:

* Not completing 18 years of age
* not willing to volunteer to study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: consists of volunteer healthy individuals.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
6 Minute Pegboard and Ring Test | A total of one measurements will be made at 1-week
  The 6-minute pegboard and ring test is used to assess upper extremity functional capacity. The patient sat in front of a perforated board with bottom pegs at shoulder level. The upper pegs are placed in the hole 20 cm above the lower pegs. 10 rings of the same size are placed on the lower pegs. The patient is asked to move as many rings as possible from the lower pegs to the upper pegs and vice versa within a 6-minute period. Pulse, blood pressure, SpO₂, dyspnea and arm fatigue detection are recorded before/after each test. Before the actual test, patients are allowed to move up and down the rings in a cycle to become familiar with the testing procedure. If the patient wants to rest during the test, he is allowed, but the stopwatch is not stopped. During the test, standard encouraging phrases are said to the patient at the end of each minute.
Immersive virtual reality version of the 6 Minute Pegboard and Ring Test | A total of two measurements will be made at 1-week intervals within 6 months.
  The classic 6-minute pegboard and ring test adapted to the virtual environment

SECONDARY OUTCOMES:
Quick Shoulder-Hand Syndromes Questionnaire | A total of two measurements will be made at 1-week intervals within 6 months
  The Quick Shoulder-Hand Syndromes Questionnaire is used to evaluate musculoskeletal physical function and symptoms of the upper extremity. The survey consists of 11 items and is scored between 0-100 points. Higher scores indicate more disability
Assessment of handgrip | A total of two measurements will be made at 1-week intervals within 6 months
  Hand grip strength was evaluated with a dynamometer. The best score was recorded by taking 3 measurements separately for left and right hand.
9 Hole Peg Test | A total of two measurements will be made at 1-week intervals within 6 months
  The 9-hole peg test is a standardised test that measures fine dexterity against time. It is a simple test and is a valid and reliable method of assessment. Both hands are tested in the assessment

CONTACTS AND LOCATIONS:
Overall Officials: Çağtay MADEN, PhD, Principal Investigator — Gaziantep İslamic Science and Technology University
Locations (1):
- Gaziantep İslamic Science and Technology University, Gaziantep, Şahinbey, Turkey (Türkiye)